CLINICAL TRIAL: NCT00089492
Title: A Phase II Open-label, Randomized, Active-controlled Study Comparing the Efficacy and Safety of Once Daily Enfuvirtide Dosing Versus the Currently Recommended Twice Daily Dosing in HIV-1 Infected Treatment-experienced Patients.
Brief Title: A Study Comparing the Efficacy and Safety of Once-Daily Fuzeon (Enfuvirtide) Dosing Versus the Currently Recommended Twice-Daily Dosing in Human Immunodeficiency Virus-Type 1 (HIV-1) Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV17658
Record Dates: First submitted 2004-08-05; First posted 2004-08-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Optimized Background ARVs; Drug: enfuvirtide [Fuzeon]
- 2 (Active Comparator)
  Interventions: Drug: Optimized Background ARVs; Drug: enfuvirtide [Fuzeon]

INTERVENTIONS:
Drug: Optimized Background ARVs — As prescribed
Drug: enfuvirtide [Fuzeon] — 180mg sc once daily for 48 weeks
  Arms: 1
Drug: enfuvirtide [Fuzeon] — 90mg sc bid for 48 weeks
  Arms: 2

SUMMARY:
This study will assess the safety and efficacy of once-daily administration of Fuzeon compared with twice-daily administration in HIV-1 infected patients who have received prior treatment. Patients will also receive an optimized treatment consisting of antiretroviral (ARV) therapy as determined by the treating physician. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults or adolescents >=16 years of age;
* HIV-1 RNA >=5000 copies/mL;
* prior experience or documented resistance to each of the 3 currently available classes of ARV drugs (nucleoside reverse transcriptase inhibitors, non-nucleoside reverse transcriptase inhibitors, and protease inhibitors).

Exclusion Criteria:

* history of prior use of Fuzeon or T-1249;
* female patients who are pregnant or breastfeeding, or who plan to become pregnant during the study;
* current severe illness;
* currently taking drugs affecting the immune system, HIV vaccine, or investigational agents for any conditions other than HIV/AIDS.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Viral load.\n\n | Week 48

SECONDARY OUTCOMES:
CD4 lymphocyte count. | Week 48
AEs, laboratory abnormalities, local injection site reactions, AIDS-defining events.\n | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (19):
  - Hobson City, Alabama
  - Fountain Valley, California
  - Los Angeles, California
  - Denver, Colorado
  - Bradenton, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Atlanta, Georgia
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Union, New Jersey
  - Albany, New York
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Houston, Texas
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Puerto Rico (2):
  - Ponce
  - San Juan

REFERENCES:
- [Derived] Wright D, Rodriguez A, Godofsky E, Walmsley S, Labriola-Tompkins E, Donatacci L, Shikhman A, Tucker E, Chiu YY, Chung J, Rowell L, Demasi R, Graham N, Salgo M. Efficacy and safety of 48 weeks of enfuvirtide 180 mg once-daily dosing versus 90 mg twice-daily dosing in HIV-infected patients. HIV Clin Trials. 2008 Mar-Apr;9(2):73-82. doi: 10.1310/hct0902-73. PMID 18474492